CLINICAL TRIAL: NCT07292727
Title: Effect of Virtual Reality on Pain and Anxiety During Chemotherapy Session in Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hanaa Hassanin Shehata Hassan, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005460
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional care group (Active Comparator): This group includes patients suffering from pain and anxiety. Patients will receive their traditional care at every chemotherapy session
  Interventions: Other: traditional care
- Virtual reality group (Experimental): This group includes patients suffered from pain and anxiety. The patients received their traditional care in addition to a fully immersive Head-Mounted Display virtual reality.
  Interventions: Other: traditional care; Other: Virtual reality

INTERVENTIONS:
Other: traditional care — Patients will take their prescribed medications from their physician and will continue their traditional activities during the intervention period, including reading, watching television, or visiting with guests.
Other: Virtual reality — The patients will receive their traditional care in addition to a fully immersive Head-Mounted Display virtual reality (Oculus meta Quest virtual reality (VR) headset with hand controller ) for 30 minutes, starting from the patient's second chemotherapy session and last for 3 sessions.
  Arms: Virtual reality group

SUMMARY:
This study will be conducted to determine the effect of virtual reality exercise on pain and anxiety in breast cancer patients during chemotherapy treatment

DETAILED DESCRIPTION:
Many breast cancer survivors experience physical and psychological symptoms (such as pain, fatigue, depression, anxiety, and lymphedema); functional deficits (such as reduced shoulder range of motion and cognitive impairment); emotional problems (such as fatigue, pain, anxiety, and depression); and other complications such as bleeding, effusion, and flap necrosis. Side effects from breast cancer or treatment can have a significant impact on the quality of life (QoL) of breast cancer survivors.

Anxiety is present in about 10% of people during chemotherapy, while one-third of people with depression also show clinically significant anxiety states.

Pain occurs in 90% of patients treated with chemotherapy. Pain includes that produced by the neurotoxic action of antiblastic drugs, mechanical pressure of the tumor mass, metastases and pain in the phantom limb.

Over the last two decades, virtual reality (VR), has shown efficacy as a distraction tool to alleviate pain and distress during medical procedures. The need of this study is developed from the lack in the quantitative knowledge and information in the published studies about the effect of virtual reality on pain and anxiety in cancer patient during chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with breast cancer.
* Patients who suffered from pain.
* Patient who suffered from anxiety.
* Patients who received chemo since 1cycle (session).
* Patients who received the same type of chemotherapy.
* Patients who are not suffer from anxiety disorders before chemotherapy.
* Patient who received chemotherapy for the first time in their treatment.

Exclusion Criteria:

The potential participants will be excluded if they have one of the following criteria:

* injuries to the face or head
* Hand Injuries.
* Cognitive impairment
* A history of severe motion sickness
* Mental health problems.
* Visual and auditory problems.
* Radiotherapy
* A history of skull structure or cervical spine abnormalities that may complicate the use of VR devices.
* A history of epilepsy, seizures, vertigo.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain intensity | 6 weeks
  Numerical rating scale (NRS) will be used to assess pain intensity. Pain levels will assess after the start of chemo infusion and immediately after intervention of VR for each session. The type of pain measured refers to any painful symptomatology that a cancer patient undergoing chemotherapy may experience. NRS score: "no pain = 0," "mild pain = 1-4," "moderate pain = 5-6," and "severe pain = 7-10."
Assessment of anxiety | 6 weeks
  Hamilton anxiety scale (HAM-A) will be used to assess anxiety level. The HAM-A entails 14 items, each categorized by a series of symptoms, and measures mental agitation and psychological distress, as well as anxiety-related physical complaints. The responses on the scale were measured on a 5-point Likert scale: 0 (symptoms not present), 1 (mild symptoms), 2 (moderate symptoms), 3 (severe symptoms) and 4 (very severe symptoms). The total score was calculated by summation of the 14 items. Each item is scored on a scale of 0 (not present) to 4(severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Khalifa, Professor, Study Director — Sohag University; Mohamed KhallafK, Professor, Study Chair — Cairo University
Locations (1):
- Hanaa Hassanin Shehata, Sohag, Egypt